CLINICAL TRIAL: NCT06163157
Title: Investigation of the Effectiveness of Connective Tissue Massage in Individuals With Erectile Dysfunction Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bitlis Eren University (Other)
Responsible Party: Principal Investigator, Mesut Arslan, Assistant Professor, Bitlis Eren University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ED-CTM
Record Dates: First submitted 2023-11-20; First posted 2023-12-08 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Erectile Dysfunction
Keywords: Erectile dysfunction; Connective tissue massage
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control roup (No Intervention): The control group will receive standard treatment (lifestyle recommendations).
- CTM group (Experimental): In addition to the standard treatment, connective tissue massage will be applied to the CTM group.
  Interventions: Other: Connective tissue massage(CTM)

INTERVENTIONS:
Other: Connective tissue massage(CTM) — CTM will be applied by a trained physiotherapist for 3 days/week for 4 weeks. Application time will be approximately 15-20 minutes.
  Arms: CTM group

SUMMARY:
In this study, it is planned to investigate the effect of connective tissue massage on symptom severity, autonomic functions, psychological state and quality of life in individuals with erectile dysfunction symptoms.

DETAILED DESCRIPTION:
The most common sexual dysfunctions in men include erectile dysfunction and premature ejaculation. Erectile dysfunction (ED) is defined as the inability to achieve and maintain the penile erection necessary for sexual intercourse for at least 6 months.The prevalence of ED generally varies between 37.2%-48.6%.

There are various treatment methods used in individuals with ED symptoms. While urologists use oral phosphodiesterase-5 inhibitor drugs (such as sildenafil and vardenafil) as the first step, intracavernosal papaverine or alprostadil injections and vacuum devices may be preferred afterwards. When these treatments are inadequate, penile prostheses can be used. In addition, various physiotherapy techniques such as pelvic floor muscle training, electrical stimulation, massage and aerobic exercises are also recommended for these individuals.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects aged 20-65 years with ED complaints for at least 6 months will be included in the study. In addition, sexually active individuals will be included in the study

Exclusion Criteria:

* Patients with diabetes and renal diseases, uncontrolled hypertension, priapism, pacemaker users, history of psychiatric or psychological illness, skin lesions/ulcer in the penis or lumbosacral region, and patients who are unable to cooperate will be excluded.

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-12-21 (Actual); Primary Completion 2024-12-21 (Actual); Study Completion 2024-12-21 (Actual)

PRIMARY OUTCOMES:
The International Index of Erectile Function (IIEF-5) | Change from baseline at 4 weeks
  İt is a 5-question questionnaire used to assess erectile dysfunction. Patients' answers to each question are scored between 1 and 5. A total score above 21 indicates normal erectile function, while a score of 21 and below indicates ED. According to the total score obtained from the scale, ED is divided into 4 categories. Severe (1-7), moderate (8-11), moderate to mild (12-16), mild (17-21) and no ED (22-25).
Composite Autonomic Symptom Score (COMPASS 31) | Change from baseline at 4 weeks
  İt is a 31-question questionnaire that assesses autonomic symptoms in 6 different areas: orthostatic intolerance, vasomotor, secretomotor, gastrointestinal, bladder function and pupillomotor. Survey score varies between 0-100 points. A high score on the questionnaire indicates the presence and severity of autonomic dysfunction.

SECONDARY OUTCOMES:
Depression Anxiety Stress Scale (DASS-21) | Change from baseline at 4 weeks
  It evaluates the condition of the individual in the last week. It is a 21-question questionnaire consisting of 3 subscales: depression, anxiety and stress. Survey score varies between 0-63 points. A high score on the questionnaire indicates the presence and severity of depression, anxiety and stress.
Quality of Life Questionnaire (SF-36) | Change from baseline at 4 weeks
  It is a 36-question questionnaire consisting of 8 subscales including physical function, physical role, emotional role, pain, vitality, general health and mental health. Survey score varies between 0-100 points. A high score obtained from the questionnaire indicates that the individual has a good quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Bitlis Eren University, Bitlis, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No